CLINICAL TRIAL: NCT01299714
Title: Community Awareness, Resources and Education (CARE II): Project 3
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Michigan (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Electra Paskett, Marion N. Rowley Professor of Cancer Research and Director-Division of Cancer Prevention and Control, Ohio State University
Other Study IDs: OSU-10096; P50CA105632 (NIH); OSU-10096 (Other: OSU Comprehensive Cancer Center)
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Uterine Cervical Cancer
Keywords: Human Papilloma Virus; vaccine; stress; cervical cancer; GARDASIL
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, Pap specimen, cervical specimen for HPV analysis, oral rinse specimen, saliva specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Researchers at The Ohio State University and the University of Michigan are working together to understand cancer of the cervix. One of the areas they are studying is how stress you may experience in your life effects the way you respond to GARDASIL®. GARDASIL® is a vaccine approved by the Food and Drug Administration (FDA) to prevent some types of Human Papillomavirus (HPV) infection which can cause cancer of the cervix. Participants are being recruited from the Appalachian region of Ohio.

DETAILED DESCRIPTION:
A quadrivalent HPV 6, 11, 16, 18 vaccine (GARDASIL®) has been approved for use among women age 9-26 years to prevent cervical/vaginal/vulvar cancer and genital warts. The efficacy of the vaccine has been demonstrated in clinical trial settings, but the effectiveness of this vaccine has not been tested in clinical practice settings. Patients experiencing greater stress have a reduced capacity to mount an immune response to other types of vaccine. The same phenomenon is likely to exist for Gardasil, but there are no data. The impact of psychological stress on the immune response to a vaccine is proposed to act via health behaviors (multiple lifetime sexual partners, never using condoms, prior abnormal Pap smear, smoking, and HPV infection) or by direct dysregulation of the immune system. We have found higher rates of cervical HPV in Appalachian Ohio women, higher rates of abnormal cervical cytology, and very high rates of psychological stress compared to urban and suburban women. The goal of this study is to determine if, in women age 18-26 years given GARDASIL® vaccine, serum HPV 6/11/16/18 antibody response is altered by stress. This will be accomplished by a study of 432 women age 18-26 years who report full range of life stressors recruited from Appalachian Ohio. All participants will receive the GARDASIL® vaccine at baseline, two months, and six months. Prior to vaccination questionnaire data related to HPV exposure risk behaviors and psychological stressors will be collected. Cervical samples will be collected for cytology and HPV testing. Serum samples will be collected for HPV 6, 11, 16 and 18 antibody assays at baseline and month 12. The questionnaire data and serum samples will be repeated at 12 months. The primary outcome measure is the difference in serum antibodies to HPV 6, 11, 16 and 18 at baseline and month 12. The variables of interest are perceived stress, sexual behaviors, socioeconomic status, access to health care (health insurance yes/no), smoking, Appalachian self-identity, HPV cervical status at baseline, and past history abnormal cervical cytology, as proposed in a psychoneuroimmunology model. In this model, Appalachian Self-Identity, socioeconomic status, loneliness, health care access, and coping are proposed to contribute to a woman's perceived stress. The impact of perceived stress on immune response to Gardasil vaccination can be by health behaviors such as multiple lifetime sexual partners (>4), never using condoms, prior abnormal Pap smear, smoking, and HPV status at the time of vaccination. Perceived stress can have a direct physiologic impact on the immune response by creating immune dysregulation as measured by increased EBV VCA-IgG titers. Depressive symptoms can mediate the impact of perceived stress on immune function. If psychological stress is found to modulate the immune response to GARDASIL®, then we can determine if the modulation reduces the clinical effectiveness of the vaccine and examine methods to limit the impact of stress.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-26 years of age
* Resident of an Appalachian county
* Intact cervix
* Able to read and understand English
* Cognitively able to provide informed consent
* Willing to come for four clinic visits

Exclusion Criteria:

* Prior history of cervical cancer
* Prior history of a cervical lesion treated with cryotherapy or any form of surgical removal of a portion of the cervix to treat CIN
* No cervix
* Pregnant or planning to become pregnant in the next year
* History of immune disorder: auto-immune, primary immune or acquired
* Any contra-indications for the GARDASIL® vaccine series
* Taking immune suppressive medications
* Any prior exposure to an HPV vaccine of any type
* Planning to move out of the immediate area in the next year

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be female, aged 18 - 26 years, residing in an Appalachian region, with no history of HPV vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
serum antibody levels for HPV 6,11,16 and 18 | 12 months

SECONDARY OUTCOMES:
serum antibody levels for Epstein-Barr Virus (EBV) | baseline
Center for Epidemiological Studies - Depression (CES-D) Scale Score | 12 months
perceived stress | 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Mack T Ruffin, IV, MD, MPH, Principal Investigator — University of Michigan; Electra D Paskett, PhD, Study Director — Ohio State University
Locations (4):
- United States (4):
  - Athens, Ohio
  - Gallipolis, Ohio
  - Logan, Ohio
  - Pomeroy, Ohio

REFERENCES:
- See also: CARE: Project 3 Study — http://www.CAREProject3.osu.edu